CLINICAL TRIAL: NCT01089816
Title: Clinical Validation of the Point-of-Care MSD Influenza Test in Asia
Brief Title: Rapid Diagnostic Test for Influenza
Status: Completed | Type: Observational
Sponsor: Meso Scale Diagnostics, LLC. (Industry)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency)
Responsible Party: Sponsor
Other Study IDs: SEA034
Record Dates: First submitted 2010-03-16; First posted 2010-03-19 (Estimated); Last update posted 2015-04-21 (Estimated); Status verified 2015-04

CONDITIONS: Influenza
Keywords: Influenza infections; Orthomyxoviridae infections; Influenza Human
MeSH Terms: conditions — Influenza, Human; Orthomyxoviridae Infections

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Viral transport media containing nasal swab extract.
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- All: Anyone presenting with influenza-like-illness
  Interventions: Biological: Local/Regional Public Health Notification

INTERVENTIONS:
Biological: Local/Regional Public Health Notification — For any H5 positive results, notification of the result to the site's local/regional public health authorities.

SUMMARY:
The primary objective of this study is to evaluate the performance of the MSD® Influenza Test in detecting influenza A and influenza B in subjects presenting with influenza-like-illness (ILI).

DETAILED DESCRIPTION:
This is a multicenter, prospective study to evaluate the performance of the MSD Influenza Test for the detection and differentiation of influenza A (including A/H1, A/H3, and A/H5 subtypes) and influenza B. Nasal swabs from subjects presenting at the clinical care facility with ILI will be collected and tested on the MSD Influenza Test. Results from the Test will be compared to results obtained from viral culture performed on a second nasal swab at a reference laboratory.

ELIGIBILITY:
Inclusion Criteria:

* Any subject (all ages) presenting with ILI (defined as fever [subjective or documented] and cough or sore throat), and suspected of having influenza.
* Subject (parent, guardian, or authorized legal representative) gives informed consent to the study, and provides signed authorization for use and disclosure of protected health information.

Exclusion Criteria:

* Subjects who had prior nasal wash/aspirate or nasopharyngeal wash/aspirate specimens collected for routine health-care purposes within the same suspected influenza infection episode.
* Unable to collect nasal and throat swab.
* Severely ill patient without a family relative to provide informed consent.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Individuals visiting a health care facility.
Sampling Method: Non-Probability Sample
Enrollment: 569 (Actual)
Dates: Start 2010-03; Primary Completion 2010-08 (Actual); Study Completion 2010-10 (Actual)

PRIMARY OUTCOMES:
To determine the sensitivity and specificity of influenza A and B, and subtypes A/H1 and A/H3 with nasal and throat specimens for the MSD Influenza test as compared to cell culture and sequencing in a cross-section of the general population | 4 months

SECONDARY OUTCOMES:
To determine the specificity of influenza subtype A/H5 in nasal and throat specimens for the MSD Influenza test as compared to cell culture and sequencing in a cross section of the general population. | 4 months

CONTACTS AND LOCATIONS:
Overall Officials: Jacqueline Perodin, PhD, CCRP, Study Director — Meso Scale Diagnostics
Locations (4):
- Vietnam (4):
  - National Hospital of Pediatrics, Hà Nội
  - Children's Hospital #2, Ho Chi Minh City
  - Children's Hospital 1, Ho Chi Minh City
  - Hospital for Tropical Diseases, Ho Chi Minh City